CLINICAL TRIAL: NCT02955784
Title: Sinasprite: A Pilot Feasibility Study of a Casual Game for Primary Care Patients With Mild Stress, Anxiety or Depression
Brief Title: Sinasprite: A Pilot Feasibility Study for Patients With Anxiety or Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215019
Record Dates: First submitted 2015-01-06; First posted 2016-11-04 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Stress; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sinasprite Mobile App (Experimental): Mobile App
  Interventions: Device: Sinasprite Mobile App

INTERVENTIONS:
Device: Sinasprite Mobile App — Mobile App

SUMMARY:
The investigators are proposing a prospective one-arm cohort study testing the feasibility of a game designed to improve symptoms in adults with mild levels of stress, depression, and anxiety. The study will take place at Madigan Army Medical Center. Primary outcomes include usage data including time, frequency and duration of app use, participant satisfaction with the game, and comments and suggestions regarding participants' experiences using the Sinasprite game over a 12-week period. Participants will download Litesprite's game, Sinasprite, onto their personal smartphone. Elements of cognitive-behavioral therapies like cognitive strategies, diaphragmatic breathing, and visualization are embedded in the game enabling participants to learn to achieve the desired healthy habits. The game's goal is to help Socks the Fox become a Zen Master. Over six weeks, players help Socks to progress by describing and categorizing their concerns, entrusting Socks to "hold" these concerns, and engaging in bonding activities with Socks, such as fishing and meditation. The investigators currently have a prototype and have been told by insurance firms, providers, and self-funded employers that they need to see validated results from a pilot study that shows feasibility with subjects in the target audience before they can consider a commercial roll out. Participants will complete questions related to mood, stress, and well-being at baseline, 6 weeks, and 12 weeks. Data will be evaluated in real-time and reports of participant progress will be provided to the participant's provider, with the participant's consent. Data and feedback from this pilot study will be used to update the design and inform the technical development team to further refine the game experience in preparation for a larger randomized controlled trial evaluating the effectiveness of Sinasprite.

DETAILED DESCRIPTION:
In the U.S. anxiety disorders cost over $55 billion, and major depression is second only to back and neck pain for having the greatest impact on disability days at 386.6 million days/year. Primary care providers (PCPs) are overwhelmingly responsible for screening and treating their patients for behavioral health conditions such as depression and anxiety, and approximately 70-80% of antidepressants are prescribed in primary care. Nearly 17% of the population will experience depression at some point in their lifetime, but of those treated for depression in the primary care setting, only 20-40% show substantial improvement over 12 months. Insurance companies spend $1 trillion annually on behavioral health conditions. $250 billion is spent on our target segment - those with high stress or mild to moderate depression/anxiety, but no serious mental illness requiring intensive or inpatient treatment. These populations have significantly adopted and use mobile technologies for health purposes. Current solutions, like AppsRx, ORCAS, or SuperBetter, are clinically-focused or, at best, use game elements as opposed to a full gaming experience and do not target payers or hospitals. LinkedWellness has a true gaming experience for anxiety/depression, but their target audience is solely focused on teens. None of these incorporate the player's social networks, biosensors, collect information from the phone, or provide predictive insights. Therefore, tools to enhance management of these patients in a primary care setting, such as the casual health-related game Sinasprite, may improve treatment of difficult-to-manage behavioral health conditions. The investigators are proposing a prospective one-arm cohort study testing the feasibility of a game designed to improve symptoms in adults with mild levels of stress, depression, and anxiety. The study will take place at Madigan Army Medical Center. Primary outcomes include usage data including time, frequency and duration of app use, participant satisfaction with the game, and comments and suggestions regarding participants' experiences using the Sinasprite game over a 12-week period. Participants will download Litesprite's game, Sinasprite, onto their personal smartphone. Elements of cognitive-behavioral therapies like cognitive strategies, diaphragmatic breathing, and visualization are embedded in the game enabling players to learn to achieve the desired healthy habits. The game's goal is to help Socks the Fox become a Zen Master. Over six weeks, players help Socks to progress by describing and categorizing their concerns, entrusting Socks to "hold" these concerns, and engaging in bonding activities with Socks, such as fishing and meditation. The investigators currently have a prototype and have been told by insurance firms, providers, and self-funded employers that they need to see validated results from a pilot study that shows feasibility with subjects in the target audience before they can consider a commercial roll out. Participants will complete questions related to mood, stress, and well-being at baseline, 6 weeks, and 12 weeks. Data will be evaluated in real-time and reports of participant progress will be provided to the participant's provider, with the participant's consent. Data and feedback from this pilot study will be used to update the design and inform the technical development team to further refine the game experience in preparation for a larger randomized controlled trial evaluating the effectiveness of Sinasprite.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Eligible to receive care at a MHS clinic
3. English-speaking
4. In possession of a personal smartphone capable of downloading the Sinasprite application for use during the study
5. Self-reported PHQ-9 score ≤ 10 and no self-reported suicidal or homicidal ideation
6. Self-reported GAD-7 score ≤ 10 and no self-reported suicidal or homicidal ideation
7. No change in antidepressant or antianxiety medication and/or dosage in past 3 months

Exclusion Criteria:

1. Under 18 years of age
2. English insufficient to interact with the game or complete assessments
3. Residing in an institution or other living situation where health care decisions are not made by the participant (e.g., hospitalized, prisoners, people living in a rehabilitation facility)
4. Self-reported PHQ-9 score > 10 or self-reported suicidal or homicidal ideation
5. Self-reported GAD-7 score > 10 or self-reported suicidal or homicidal ideation
6. Change in antidepressant or antianxiety medication and/or dosage in past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction. These data will be collected via questionnaire at the end of the study only | 12 wks
  Data is via a standardized satisfaction questionnaire developed by the authors that is a mixture of open ended and likert scale questions on satisfaction with the app.

SECONDARY OUTCOMES:
Measure of perceived stress (PSS) | Pre/post (0, 6 and 12 wks)
  Participants will complete the 10 item perceived stress scale (PSS validated questionnaire) at 0, 6 and 12 wks.
Quality of life (LiSAT-9) | Pre/post (0, 6 and 12 wks)
  Participants will complete the LiSAT-9 validated questionnaire at 0, 6, and 12 weeks to assess their quality of life during the study.
Symptom reports: measure of depression symptoms (PHQ-9 score) | Pre/post (0, 6, and 12 wks)
  Participants will complete the 9 item PHQ-9 validated questionnaire at 0, 6, and 12 wks to assess participant symptoms of self-reported depression during the study.
Symptom reports: measure of anxiety symptoms (GAD-7 score) | Pre/post (0, 6, and 12 wks)
  Participants will complete the 7 item GAD-7 validated questionnaire at 0, 6, and 12 wks to assess participant symptoms of self-reported anxiety during the study.
Measure of coping self-efficacy (CSE) questionnaire | Pre/post (0, 6 and 12 wks)
  Participants will complete the 26 item coping self-efficacy (CSE) validated questionnaire at 0, 6 and 12 wks to assess their coping self-efficacy during the study.
App daily usage (minutes/day) | 12 wks
  Time (minutes per day) app was used
App frequency usage (days/week) | 12 wks
  Frequency (days/week) app was used
App duration of usage (total weeks) | 12 wks
  Weeks app was used

CONTACTS AND LOCATIONS:
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study still in data collection process